CLINICAL TRIAL: NCT01787383
Title: A Simultaneous Treatment Regimen Compared to a Sequential Treatment Regimen With Ingenol Mebutate Gel 0.015% and 0.05% of Two Areas With Actinic Keratosis on Face/Scalp and Trunk/Extremities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP0041-64; 2012-002863-88 (EudraCT Number)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2021-05

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Ingenol mebutate gel
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ingenol mebutate gel 0.05 % (Active Comparator)
  Interventions: Drug: Ingenol mebutate gel 0.05 %; Drug: Ingenol mebutate gel 0.015 %
- Ingenol mebutate gel 0.015 % (Active Comparator)
  Interventions: Drug: Ingenol mebutate gel 0.05 %; Drug: Ingenol mebutate gel 0.015 %

INTERVENTIONS:
Drug: Ingenol mebutate gel 0.05 % — Ingenol mebutate gel 0.05 % (Picato®) on trunk/extremities either applied simultaneously or sequentially
  Other Names: Picato®
Drug: Ingenol mebutate gel 0.015 % — Ingenol mebutate gel 0.015 % (Picato®) on face/scalp either applied simultaneously or sequentially
  Other Names: Picato®

SUMMARY:
The purpose of this trial is to evaluate the safety of a simultaneous treatment regimen compared to a sequential treatment regimen when two separate areas with AKs (one located on face/scalp and the other located on trunk/ extremities) are treated with ingenol mebutate gel

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide informed consent
* Subjects with 4 to 8 clinically typical, visible and discrete AKs within a contiguous 25 cm2 treatment area on face or scalp
* Subjects with 4 to 8 clinically typical, visible and discrete AKs within a contiguous 25 cm2 treatment area on trunk or extremities
* Subjects at least 18 years of age
* Female subjects must be of either:

  1. Non-childbearing potential, i.e. post-menopausal or have a confirmed clinical history of sterility (e.g. the subject is without a uterus) or,
  2. Childbearing potential, provided there is a confirmed negative urine pregnancy test prior to trial treatment, to rule out pregnancy.
* Female subjects of childbearing potential must be willing to use effective contraception at trial entry and until completion.

Exclusion Criteria:

* Location of the selected treatment areas:

  * on the periorbital skin
  * within 5 cm of an incompletely healed wound
  * within 10 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC)
* Prior treatment with ingenol mebutate gel on face/scalp and on trunk/extremities
* Lesions in the selected treatment areas that have:

  * atypical clinical appearance (and/or,
  * recalcitrant disease
* History or evidence of skin conditions other than the trial indication that would interfere with the evaluation of the trial medication
* Use of cosmetic or therapeutic products and procedures which could interfere with the assessments of the selected treatment areas
* Clinical diagnosis/history or evidence of any medical condition that would expose a subject to an undue risk of a significant AE or interfere with assessments of safety and efficacy during the course of the trial, as determined by the investigator's clinical judgment.
* Anticipated need for hospitalisation or out-patient surgery during the first 15 days after the first trial medication application.
* Known sensitivity or allergy to any of the ingredients in ingenol mebutate gel
* Presence of sunburn within the selected treatment areas
* Current enrolment or participation in an investigational clinical trial within 30 days of entry into this trial
* Subjects previously randomised in the trial
* Female subjects who are breastfeeding
* In the opinion of the investigator, the subject is unlikely to comply with the Clinical Study Protocol

Prohibited Therapies and/or Medications within 2 weeks prior to Visit 1:

* Cosmetic or therapeutic procedures within 2 cm of the selected treatment areas
* Use of topical keratolytic therapeutic products within 2 cm of the selected treatment areas
* Use of topical medicated creams, ointments, lotions, gels, foams or sprays including topical steroids : within 2 cm of the selected treatment areas; artificial tanners: within 5 cm of the selected treatment areas

Prohibited Therapies and/or Medications: within 4 weeks prior to Visit 1:

* Treatment with immunomodulators, cytotoxic drugs or interferon/interferon inducers
* Treatment with systemic medications that suppress the immune system
* Treatment/therapy with ultraviolet light A (UVA) or ultraviolet light B (UVB)

Prohibited Therapies and/or Medications within 8 weeks prior to Visit 1:

- Treatment with 5-fluorouracil (5-FU), imiquimod, topical diclofenac sodium, or photodynamic therapy within 2 cm of the selected treatment areas.

Prohibited Therapies and/or Medications within 6 months prior to Visit 1:

- Use of systemic retinoids or biologic/monoclonal antibody therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- Clinica Dermatologica dell'Università di Modena e Reggio Emilia, Modena, Italy

REFERENCES:
- [Derived] Pellacani G, Peris K, Guillen C, Clonier F, Larsson T, Venkata R, Puig S. A randomized trial comparing simultaneous vs. sequential field treatment of actinic keratosis with ingenol mebutate on two separate areas of the head and body. J Eur Acad Dermatol Venereol. 2015 Nov;29(11):2192-8. doi: 10.1111/jdv.13211. Epub 2015 Aug 24. PMID 26300464

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the clinical study protocol 200 subjects were planned to be enrolled and 199 subjects were actually enrolled and randomised.
Groups:
- Ingenol Mebutate Gel Simultaneous Treatment: Ingenol mebutate gel in 2 doses (0.015 %: and 0.05 %) were applied simultaneously: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities.
- Ingenol Mebutate Gel Sequential Treatment: Ingenol mebutate gel in 2 doses (0.015 %: and 0.05 %) were applied sequentially: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities.
Period: Overall Study
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment
Started | 101 | 98
Completed | 92 | 76
Not Completed | 9 | 22

BASELINE CHARACTERISTICS:
Groups:
- Ingenol Mebutate Gel Simultaneous Treatment: Ingenol mebutate gel 0.05 %: Ingenol mebutate gel 0.05 % (Picato®) on trunk/extremities applied simultaneously
  Ingenol mebutate gel 0.015 %: Ingenol mebutate gel 0.015 % (Picato®) on face/scalp applied simultaneously
- Ingenol Mebutate Gel Sequential Treatment: Ingenol mebutate gel 0.05 %: Ingenol mebutate gel 0.05 % (Picato®) on trunk/extremities applied sequentially
  Ingenol mebutate gel 0.015 %: Ingenol mebutate gel 0.015 % (Picato®) on face/scalp applied sequentially
- Total: Total of all reporting groups
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment | Total
Number analyzed (Participants) | 101 | 98 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 9 | 21
  >=65 years | 89 | 89 | 178
Age, Continuous [Mean (Full Range); unit: years] | 74.4 [43 to 94] | 74.5 [48 to 92] | 74.5 [43 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 88 | 80 | 168
Region of Enrollment [Number; unit: participants]
  Italy | 63 | 61 | 124
  Spain | 38 | 37 | 75

OUTCOME MEASURES:

1. Primary Outcome: Composite Local Skin Reaction (LSR) Score 3 Days After Treatment of Each Selected Treatment Area
Description: Composite Local Skin Reaction (LSR) score 3 days after treatment of each selected treatment area in both treatment groups (simultaneous or sequential). The composite LSR score (0 to 24), reflecting the sum of the individual LSR grades (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration, grade 0 to 4), was calculated for each selected treatment area at each visit.The composite LSR score ranges from 0 (best possible outcome) to 24 (worst possible outcome). Both affected areas were calculated together "Per Arm". Each subject could contribute with up to 2 values (1 for each treated area).
Time Frame: 3 days after treatment of each selected treatment area
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment
Number analyzed (Participants) | 101 | 98
units on a scale | 10.4 (5.1) | 9.7 (4.5)
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel Simultaneous Treatment vs Ingenol Mebutate Gel Sequential Treatment; Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Complete Clearance of AKs in Each Separate Treatment Area 8 Weeks After Treatment
Description: Complete clearance of Actinic Keratosis lesions (AKs) analysed in each separate treatment area and presented by treatment regimen given as "percentage of participants" with complete AK clearance. Each subject could contribute with up to 2 values (1 for each treated area). Both affected areas were calculated together "Per Arm" (e.g. "averaged").
Time Frame: 8 weeks after treatment
Measure: Number; unit: percentage of participants
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment
Number analyzed (Participants) | 101 | 98
percentage of participants | 52.7 | 46.9
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel Simultaneous Treatment vs Ingenol Mebutate Gel Sequential Treatment; Test type: Superiority or Other; p = 0.34, Regression, Logistic

3. Secondary Outcome: Partial Clearance of AKs in Each Separate Treatment Area 8 Weeks After Treatment
Description: Partial clearance of Actinic Keratosis lesions (AKs) defined as 75% or greater reduction in Actinic Keratosis lesions (AKs) from start of treatment to 8 weeks after treatment, was analysed in each separate treatment area and presented by treatment regimen given as "percentage of participatns" with complete AK clearance. Each subject could contribute with up to 2 values (1 for each treated area). Both affected areas were calculated together "Per Arm" (e.g. "averaged").
Time Frame: 8 weeks after treatment
Measure: Number; unit: percentage of participants
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment
Number analyzed (Participants) | 101 | 98
percentage of participants | 76.6 | 68.1
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel Simultaneous Treatment vs Ingenol Mebutate Gel Sequential Treatment; Test type: Superiority or Other; p = 0.088, Regression, Logistic

4. Secondary Outcome: Percent Reduction in Number of AKs in Each Separate Treatment Area 8 Weeks After Treatment
Description: Percent reduction in number of Actinic Keratosis lesions (AKs) analysed for each separate treatment area and presented by treatment regimen. Each subject could contribute with up to 2 values (1 for each treated area). Both affected areas were calculated together "Per Arm" (e.g. "averaged").
Time Frame: 8 weeks after treatment
Measure: Mean (Standard Deviation); unit: percentage reduction in number of AKs
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment
Number analyzed (Participants) | 101 | 98
percentage reduction in number of AKs | 83.4 (22.0) | 79.1 (26.7)
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel Simultaneous Treatment vs Ingenol Mebutate Gel Sequential Treatment; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Effectiveness Satisfaction Questionnaire for Medication (TSQM)
Description: Effectiveness TSQM After a Treatment Cycle of 8 Weeks. Measurement of the perceived effectiveness of medication, ranging from 0 (worst possible outcome) to 100 (best possible outcome).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ingenol Mebutate Gel Simultaneous Treatment: Ingenol mebutate gel in 2 doses (0.015 %: and 0.05 %) were applied simultaneously: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities. The Effectiveness TSQM compliance was lower than the number of randomised subjects.
- Ingenol Mebutate Gel Sequential Treatment: Ingenol mebutate gel in 2 doses (0.015 %: and 0.05 %) were applied sequentially: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities. The Effectiveness TSQM compliance was lower than the number of randomised subjects.
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment
Number analyzed (Participants) | 90 | 73
units on a scale | 63.1 (23.4) | 66.4 (21.4)
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel Simultaneous Treatment vs Ingenol Mebutate Gel Sequential Treatment; Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Side Effects TSQM
Description: Side Effects TSQM After a Treatment Cycle of 8 Weeks. Measurement of the perceived side effects of medication, ranging from 0 (worst possible outcome) to 100 (best possible outcome).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ingenol Mebutate Gel Simultaneous Treatment: Ingenol mebutate gel in 2 doses (0.015 %: and 0.05 %) were applied simultaneously: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities. The Side EffectsTSQM compliance was lower than the number of randomised subjects.
- Ingenol Mebutate Gel Sequential Treatment: Ingenol mebutate gel in 2 doses (0.015 %: and 0.05 %) were applied sequentially: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities. The Side Effects TSQM compliance was lower than the number of randomised subjects.
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment
Number analyzed (Participants) | 90 | 73
units on a scale | 93.1 (18.4) | 96.1 (16.4)
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel Simultaneous Treatment vs Ingenol Mebutate Gel Sequential Treatment; Test type: Superiority or Other; p = 0.033, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Global Satisfaction TSQM
Description: Global Satisfaction TSQM After a Treatment Cycle of 8 Weeks. Measurement of the perceived overall satisfaction with medication, ranging from 0 (worst possible outcome) to 100 (best possible outcome).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ingenol Mebutate Gel Simultaneous Treatment: Ingenol mebutate gel in 2 doses (0.015 %: and 0.05 %) were applied simultaneously: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities. The Global Satisfaction TSQM compliance was lower than the number of randomised subjects.
- Ingenol Mebutate Gel Sequential Treatment: Ingenol mebutate gel in 2 doses (0.015 %: and 0.05 %) were applied sequentially: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities. The Global Satisfaction TSQM compliance was lower than the number of randomised subjects.
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment
Number analyzed (Participants) | 82 | 72
units on a scale | 64.6 (19.0) | 67.4 (20.3)
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel Simultaneous Treatment vs Ingenol Mebutate Gel Sequential Treatment; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Convenience TSQM
Description: Convenience TSQM After a Treatment Cycle of 8 Weeks. Measurement of the perceived convenience with medication, ranging from 0 (worst possible outcome) to 100 (best possible outcome).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ingenol Mebutate Gel Simultaneous Treatment: Ingenol mebutate gel in 2 doses (0.015 %: and 0.05 %) were applied simultaneously: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities. The Convenience TSQM compliance was lower than the number of randomised subjects.
- Ingenol Mebutate Gel Sequential Treatment: Ingenol mebutate gel in 2 doses (0.015 %: and 0.05 %) were applied sequentially: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities. The Convenience TSQM compliance was lower than the number of randomised subjects.
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment
Number analyzed (Participants) | 83 | 73
units on a scale | 73.7 (14.6) | 74.7 (18.1)
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel Simultaneous Treatment vs Ingenol Mebutate Gel Sequential Treatment; Test type: Superiority or Other; p = 0.66, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Ingenol Mebutate Gel Simultaneous Treatment: Ingenol mebutate gel in 2 doses (0.015% and 0.05%) were applied simultaneously: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities.
- Ingenol Mebutate Gel Sequential Treatment: Ingenol mebutate gel in 2 doses (0.015% and 0.05%) were applied sequentially: ingenol mebutate gel 0.015% (Picato®) was applied once daily for 3 consecutive days on on face/scalp and ingenol mebutate gel 0.05% (Picato®) was applied once daily for 2 consecutive days on trunk/extremities.
Arm/Group | Ingenol Mebutate Gel Simultaneous Treatment | Ingenol Mebutate Gel Sequential Treatment
Serious Adverse Events (participants affected / at risk) | 3/101 | 4/98
Other Adverse Events (participants affected / at risk) | 22/101 | 22/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ingenol Mebutate Gel Simultaneous Treatment (N=101) | Ingenol Mebutate Gel Sequential Treatment (N=98)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ingenol Mebutate Gel Simultaneous Treatment (N=101) | Ingenol Mebutate Gel Sequential Treatment (N=98)
Application site pruritus (General disorders) | 8 | 1
Application site pain (General disorders) | 5 | 1
Feeling cold (General disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 5 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0
Scotoma (Eye disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Application site burn (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less